CLINICAL TRIAL: NCT06771037
Title: The Use of Non-invasive Transcutaneous Auricular Neurostimulation (tAN®) in Alcohol Withdrawal Management
Brief Title: Use of tAN® in Alcohol Withdrawal Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erin Deneke (Other)
Responsible Party: Sponsor-Investigator, Erin Deneke, Senior Director of Research, Caron Treatment Centers
Organization: Caron Treatment Centers (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Caron001
Record Dates: First submitted 2025-01-02; First posted 2025-01-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Withdrawal
Keywords: Alcohol withdrawal; tAN; transcutaneous auricular neurostimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active Transcutaneous Auricular Neurostimulation (tAN) (Experimental): Transcutaneous auricular stimulation will be delivered using the Sparrow® Link in addition to treatment as usual (TAU). The Sparrow® Link will be set to the following outputs (range 0 mA - 5.0 mA, pulse width 250 µs, frequency 15 Hz at Region 1 (Vagus) and 100 Hz at Region 2 (Trigeminal). Device will be worn for 5 days.
  Interventions: Device: Transcutaneous Auricular Neurostimulation (tAN)
- Sham Transcutaneous Auricular Neurostimulation (tAN) (Sham Comparator): The Sparrow® Link will be set to the sham condition for participants in the sham group and no current will be delivered to either the inner or outer ear, but the screen will appear identical to the active group. Sham group will receive treatment as usual. Sham device will be worn for 5 days.
  Interventions: Device: Transcutaneous Auricular Neurostimulation (tAN)

INTERVENTIONS:
Device: Transcutaneous Auricular Neurostimulation (tAN) — Transcutaneous Auricular stimulation will be delivered using the Spark Biomedical Sparrow Link pulse generator with Sparrow Ascent earpieces. The Sparrow Link generator is based on FDA-cleared predicate Sparrow Ascent.

SUMMARY:
This research study is being conducted to learn if Transcutaneous Auricular Neurostimulation (tAN®) may be effective in treating alcohol withdrawal syndrome. Transcutaneous Auricular Neurostimulation (tAN®) works by delivering small electrical stimulations to the Vagus and Trigeminal nerves. This study will be conducted over the course of five days. Participants will be enrolled within 24 hours of entering treatment for alcohol withdrawal management. A total of 60 individuals will be enrolled and randomly assigned to either active (treatment with the device + treatment as usual) or sham (treatment as usual) group. Data will be collected on alcohol craving, use of comfort medications, sleep, and mood.

DETAILED DESCRIPTION:
This study will explore whether the use of a non-invasive Transcutaneous Auricular Neurostimulation (tAN®) device, Sparrow® Link, can be used to relieve symptoms of alcohol withdrawal symptoms and reduce the need for comfort medications during alcohol withdrawal management. This study will recruit 60 participants randomized to either active tAN® + Treatment as Usual (TAU) or sham tAN® + TAU, 30 participants in each arm. Data will be collected four times a day for 5 days, exploring ambient alcohol craving, mood, and sleep using Ecological Momentary Assessment (EMA; Wear-IT framework). Data for stress response, sleep and physical activity will also be collected using a fitness activity tracker (Garmin Vivosmart 4). In addition, the Clinical Institute Withdrawal Assessment, Revised (CIWA-AR) will be administered daily as well. Transcutaneous Auricular Neurostimulation has proven effective in reducing symptoms of opioid withdrawal and it is hypothesized that with the similar withdrawal symptom profile of alcohol withdrawal should prove effective in reducing symptoms of alcohol withdrawal as well.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 years old to 65 years old
2. Entering an inpatient substance use treatment program for alcohol withdrawal management.
3. Score a 27 or higher on the WHO-ASSIST V3.0
4. Is proficient in English
5. Score of a 4 or higher on the Prediction of Alcohol Withdrawal Severity Scale (PAWSS)
6. Able to provide written informed consent.
7. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. Age < 18 or > 65
2. Requires medical tapering from benzodiazepines or opioids.
3. Has a history of epileptic seizures or seizures due to alcohol withdrawal.
4. Has a cardiac pacemaker, cochlear prosthesis, neurostimulator or other device for which tAN® would be contraindicated.
5. Has abnormal ear anatomy or an ear infection is present.
6. Is pregnant.
7. Has any serious medical disease or condition which, in the judgment of the Principal Investigator or his/her designee, would make study participation unsafe, or would make intervention compliance difficult.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Institute Withdrawal Assessment Scale, Revised (CIWA-Ar) score | Baseline to end of study day 5
  Linear mixed effects models for repeated measurements will be used to evaluate the difference in changes in these primary outcomes between treatment and sham group. Mixed models take advantage of multiple measures from each individual, allowing for effects both between individuals and within each individual (e.g., across time). The CIWA-Ar is a 10-item scale measuring symptoms of alcohol withdrawal. The scores can range between 0-67. The total score is the sum of all scale items. Scores between 0-9 indicate absent to minimal withdrawal, Scores 10-19 indicate mild to moderate withdrawal and scores greater than 20 indicate severe withdrawal.
Amount of comfort medications utilized | Baseline to end of study day 5
  Medications such as ibuprofen, Librium, lorazepam, promethazine, loperamide, and acetaminophen are often used to treat alcohol withdrawal. A t-test will be utilized to compare medication usage between active and sham group.

SECONDARY OUTCOMES:
Change in ambient alcohol craving | Baseline to end of study day 5
  Change in ambient alcohol craving will be measured using a 0-100 Visual Analog Scale (VAS) delivered by smartphone using Ecological Momentary Assessment (EMA) delivered 4 times per day. EMA will be analyzed as a mixed model in the regression framework and will test effects of treatment status as between-group differences
Change in objective sleep | Baseline to end of study day 5
  Objective sleep will be measured using wrist actigraphy. Analyses of actigraphy data will examine the effect of time (i.e., study day) to identify differences across condition in the amount of sleep (i.e. minutes).
Change in subjective sleep | Baseline to end of study day 5
  Subjective sleep will be measured using EMA. Analyses of EMA data will examine the effect of time (i.e., study day) to identify differences across condition in the quality of sleep.

OTHER OUTCOMES:
Change in mood | Baseline to end of study day 5
  The impact of the Sparrow® Link treatment on mood will be primarily measured using EMA assessment and will be modeled using linear mixed models in the multilevel modeling (MLM) framework.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Deneke, Ph.D., Principal Investigator — Caron Treatment Centers
Locations (1):
- Caron Treatment Centers, Wernersville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tirado CF, Washburn SN, Covalin A, Hedenberg C, Vanderpool H, Benner C, Powell DP, McWade MA, Khodaparast N. Delivering transcutaneous auricular neurostimulation (tAN) to improve symptoms associated with opioid withdrawal: results from a prospective clinical trial. Bioelectron Med. 2022 Aug 18;8(1):12. doi: 10.1186/s42234-022-00095-x. PMID 35978394